CLINICAL TRIAL: NCT06722690
Title: Culturally Adapting Spiritually and Technologically Informed Interventions to Reduce Alcohol-Related Health Disparities Among Latinx Young Adults- Aim 3 RCT
Brief Title: ETSF for Latinx Young Adults with Alcohol Use Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Audrey Hai, Assistant Professor, Tulane University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-779; K01AA031323 (NIH)
Record Dates: First submitted 2024-11-26; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Alcohol Use Disorder (AUD)
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- eTSF (Experimental): This arm will receive the eTSF intervention. eTSF is a smartphone app intervention featuring culturally relevant content aimed at supporting Latinx young adults with alcohol use disorder in participating in 12-step groups.
  Interventions: Behavioral: eTSF
- Educational control (Active Comparator): This arm will receive educational materials on drinking problems and a list of local/online AA meetings
  Interventions: Behavioral: Educational materials

INTERVENTIONS:
Behavioral: eTSF — eTSF is a smartphone app intervention featuring culturally relevant content aimed at supporting Latinx young adults with alcohol use disorder in participating in 12-step groups.
  Arms: eTSF
Behavioral: Educational materials — Educational materials on drinking problems and a list of local/online AA meetings.
  Arms: Educational control

SUMMARY:
The goal of this clinical trial is to learn if the eTSF intervention is feasible among Latinx young adults with alcohol use disorder. The main questions it aims to answer are:

* Is eTSF feasible?
* Is eTSF effective in reducing alcohol use and increasing 12-step engagement compared to the control condition? The control condition will receive educational materials on drinking problems and a list of local/online AA meetings Participants will
* Be randomly assigned to either the eTSF condition or the control condition.
* Fill out the baseline online survey.
* Go through the eTSF app/control materials.
* And at 3 months post-baseline, fill out the follow-up online survey.

ELIGIBILITY:
Inclusion Criteria:

* YAs age 18-29
* Identify as Latinx
* Meet the Diagnostic & Statistical Manual of Mental Disorders 5th edition (DSM-5) diagnostic criteria for alcohol use disorder
* Are at least minimally motivated to change their drinking (i.e., scoring ≥3 on the University of Rhode Island Change Assessment Scale's contemplation, action, or maintenance subscales and ≤3 on the precontemplation subscale)
* Be able to provide at least one contact person to assist in tracking them for follow-up assessment

Exclusion Criteria:

* Attending any 12-step program (≥2 meetings in the past month)
* Experiencing psychotic symptoms or cognitive impairment
* In alcohol or drug treatment programs
* Taking addiction treatment medications
* Experiencing, expecting to experience, or had a history of severe/complicated withdrawal

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2027-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Recruitment feasibility | Every 4 weeks up to 2 years
  Recruitment feasibility will be measured by the number of participants screened and enrolled each month.
Randomization feasibility | From recruitment to baseline assessment up to two years
  Randomization feasibility will be measured by the number of baseline demographic variables with statistically significant group differences.
Retention/attrition feasibility | From recruitment to the end of the trial at three months.
  Retention/attrition feasibility will be measured by retention rates in each condition.
Adherence feasibility | From recruitment to the end of the trial at three months.
  Adherence feasibility will be measured by the percentage of eTSF app components used by the eTSF condition participants.
Assessment feasibility | From recruitment to the end of the trial at three months.
  Assessment feasibility will be measured by the proportion of missing data in each assessment.
Intervention credibility | From baseline to the end of treatment at three months.
  Intervention credibility will be measured using a single-item question: "On a scale from 1 to 5, where 1 indicates 'not at all' and 5 indicates 'very much,' to what extent do you believe this treatment will be beneficial for you?" Only eTSF condition participants will receive this measure.
Intervention satisfaction | From baseline to the end of treatment at three months.
  Intervention satisfaction will be measured using the mHealth Satisfaction Questionnaire, which has a total score range from 14 to 42. Higher total scores indicate greater user satisfaction with the mHealth app.
Intervention acceptability | From baseline to the end of treatment at three months.
  Acceptability will be measured using the Abbreviated Acceptability Rating Profile, which scores range from 8 to 48. Higher scores indicate greater acceptability of the intervention.
Intervention engagement | From baseline to the end of treatment at three months.
  Intervention engagement will be automatically recorded by the app during the study period and be measured in terms of app opening frequency, time spent on the app per use session (i.e., the time between opening and closing the app), most frequently used intervention component, time spent per intervention component, the completion rate of each selected component, reports of technical problems.

SECONDARY OUTCOMES:
Alcohol use | From baseline to the end of treatment at three months.
  Alcohol use will be measured using the Time-Line Follow-Back (TLFB) method-Form 90, which helps participants recall and mark days on which they used alcohol during the past 90 days.
12-Step fellowship engagement | From baseline to the end of treatment at three months.
  12-Step fellowship engagement will be measured with the Multi-Dimensional Mutual-help Activity Scale (MDMAS), which measures seven dimensions of experience (meeting attendance, meeting participation, fellowship involvement, step work, mandated attendance, affiliation, and safety). Total score ranges from 32-160 with higher scores within indicating greater engagement.

OTHER OUTCOMES:
Drinking consequences | From baseline to the end of treatment at three months.
  Drinking consequences will be measured with the Short Inventory of Problems (SIP-2R). Score ranges from 0-45 with higher scores indicating a greater frequency of experiencing problems related to substance use.
Drug use | From baseline to the end of treatment at three months.
  Drug use will be measured with the aforementioned TLFB-Form 90
Psychological distress | From baseline to the end of treatment at three months.
  Psychological distress will be assessed with the 18-item Brief Symptom Inventory. Score ranges 0-72 and higher scores indicate greater levels of psychological distress.

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be shared on the NIAAA Data Archive.